CLINICAL TRIAL: NCT04975139
Title: A Longitudinal Study to Correlate Cognitive Changes of IDH-mutant and IDH-wildtype Glioma Patients After Chemoradiotherapy With Radiation Dose to the Resting State Networks
Brief Title: Cognitive Changes of IDH-mutant and IDH-wildtype Glioma Patients After Chemoradiotherapy With Radiation Dose to the Resting State Networks
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: The Foundation for Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202006111
Record Dates: First submitted 2021-07-14; First posted 2021-07-23 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- IDH-mutant astrocytoma or oligodendroglioma: After enrollment and before beginning standard of care radiation therapy (RT), MRI will be obtained for RT planning as per standard of care (SOC), and the RS-fMRI sequences will be performed at the same time. At approximately 6 months, 2 years, 5 years, and 10 years from the completion of RT, RS-fMRIs will be performed.
  Interventions: Device: RS-fMRI
- IDH-wildtype astrocytoma: After enrollment and before beginning standard of care radiation therapy (RT), MRI will be obtained for RT planning as per standard of care (SOC), and the RS-fMRI sequences will be performed at the same time. At approximately 6 months, 2 years, 5 years, and 10 years from the completion of RT, RS-fMRIs will be performed.
  Interventions: Device: RS-fMRI
- Benign Brain Tumor: After enrollment and before beginning standard of care radiation therapy (RT), MRI will be obtained for RT planning as per standard of care (SOC), and the RS-fMRI sequences will be performed at the same time. At approximately 6 months, 2 years, 5 years, and 10 years from the completion of RT, RS-fMRIs will be performed.
  Interventions: Device: RS-fMRI

INTERVENTIONS:
Device: RS-fMRI — Advanced imaging method that can identify the spatiotemporal distribution of the intrinsic functional networks within the brain
  Other Names: Resting-state functional MRI

SUMMARY:
Neurocognitive decline after radiation therapy is one of the most concerning complication for brain tumor patients and neuro-oncologists. There are increasing technological advances in evaluating the brain's neural connections responsible for the neurocognitive processes. For example, resting-state functional MRI (RS-fMRI) is an advanced imaging method that can identify the spatiotemporal distribution of the intrinsic functional networks within the brain (also referred to as resting state networks (RSNs) without requiring specific tasks by the imaged participants. Although there is evidence that shows that avoidance of specific neural networks during radiation therapy planning can lead to improved preservation of neurocognitive function afterward, it is important to first identify the most vulnerable and clinically relevant RSNs that correspond to cognitive decline. In this study, the investigators will prospectively perform RS-fMRI and neurocognitive evaluation using the NIH Toolbox Cognitive Battery (NIHTB-CB) on patients with gliomas before and after radiation therapy to generate preliminary data on what RSNs are most vulnerable to radiation injury leading to cognitive decline. A benign brain tumor cohort will also be followed to serve as control. The investigators will also evaluate the feasibility of incorporating RS-fMRI with radiation planning software for treatment optimization.

ELIGIBILITY:
Inclusion Criteria:

* Cohort A: histological diagnosis of IDH-mutant astrocytoma or oligodendroglioma, WHO grade II-IV. IDH-mutation may be either by immunohistochemistry (IHC) or next-generation sequencing (NGS) as per routine clinical care.
* Cohort B: histological diagnosis of IDH-wildtype astrocytoma, WHO grade II-IV. IDH-wildtype status or absence of IDH-mutation may be either by IHC or NGS as per routine clinical care. The IDH-wildtype patients should have >80% probability to be alive in 6 months, and the online nomogram calculator below may be used to estimate the 6-month probability: http://cancer4.case.edu/rCalculator/rCalculator.html (Gittleman et al., 2016). The ideal patients are favorable IDH-wildtype astrocytoma patients who are expected to have prolonged survival, such as age ≤ 40 or grade 2-3 tumors.
* Cohort C: any non-infiltrative benign brain tumor histology, including but not limited to meningioma, pituitary tumor, schwannoma, craniopharngioma, hemangioblastoma, hemangiopericytoma, pineal tumor, pilocytic astrocytoma, and ganglioglioma.
* At least 18 years of age.
* Karnofsky performance status (KPS) of at least 70%
* Eligible for and planning to receive standard fractionated RT, which can be either photon-based or proton beam therapy.
* May be part of other clinical trials and can receive chemotherapy or experimental agents concurrently with or after RT as long as the other clinical trial does not exclude participation in this non-therapeutic study.
* Females of childbearing potential (defined as a female who is non-menopausal or surgically sterilized) must be willing to use an acceptable method of birth control (i.e., hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Able to understand and willing to sign an IRB-approved written informed consent document (legally authorized representative permitted).

Exclusion Criteria:

* Prior cranial RT or RT to the head and neck where potential field overlap may exist
* Gliomatosis, leptomeningeal, or metastatic involvement.
* Medical contraindication to MRI (e.g., unsafe foreign metallic implants, incompatible pacemaker, inability to lie still for long periods, severe to end-stage kidney disease or on hemodialysis).
* Require anesthesia to undergo MRI (e.g. severe claustrophobia), which would interfere with RS-fMRI acquisition and processing.
* Pregnant or breastfeeding.
* Non-English speaking, as the cognitive assessments will only be available in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen at Siteman Cancer Center at Washington University School of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2020-09-02 (Actual); Primary Completion 2033-10-31 (Estimated); Study Completion 2033-10-31 (Estimated)

PRIMARY OUTCOMES:
Change in neurocognitive scores as measured by NIH Toolbox cognitive battery tests | Prior to initiation of radiation therapy, 6 months after completion of radiation therapy, 2 years after completion of radiation therapy, 5 years after completion of radiation therapy, and 10 years after completion (estimated to be 10 years and 2 months)
  -The National Institutes of Health (NIH) has developed the National Institutes of Health Toolbox for the Assessment of Neurological and Behavior Function (NIHTB), which is a validated, normed, and multidimensional set of brief measures to assess cognitive, emotional, motor, and sensory function. The NIHTB cognitive battery (NIHTB-CB) consists of 10 tasks and can be administered in 40 min. The scores can be evaluated separately, or they can be combined into composite scores: crystallized cognition composite (reflecting the ability to access information from long-term memory and general knowledge), fluid cognition composite (reflecting the processing ability to adapt to novel environment and solve problems), and overall cognitive function composite (a combination of both crystallized and fluid scores).

SECONDARY OUTCOMES:
Change in patient reported outcomes as measured by the M.D. Anderson Symptom Inventory - Brain Tumor (MDASI-BT) | Prior to initiation of radiation therapy, 6 months after completion of radiation therapy, 2 years after completion of radiation therapy, 5 years after completion of radiation therapy, and 10 years after completion (estimated to be 10 years and 2 months)
  -The MDASI-BT is one of the most commonly used brain-specific patient-reported questionnaires on symptom burden and has been validated extensively in the adult glioma population. It can be completed in 5 minutes and allows self-reporting of symptom severity and interference with daily activities. 22 questions asking how severe are the symptoms with answers ranging from 0=not present to 10=as bad as you can imagine. 6 questions asking how the symptoms have interfered with life with answers ranging from0=did not interfere to 10=interfered completely.
Change in quality of life as measured by the Linear Analog Scale Assessment (LASA) | Prior to initiation of radiation therapy, 6 months after completion of radiation therapy, 2 years after completion of radiation therapy, 5 years after completion of radiation therapy, and 10 years after completion (estimated to be 10 years and 2 months)
  -Linear Analog Scale Assessment (LASA) is a single-item questionnaire that asks the patients to rate their overall quality of life (QOL). The LASA scale runs from 0 (as bad as it can be) to 10 (as good as it can be).
Tumor progression | Through completion of follow-up (estimated to be 10 years and 2 months)
Overall survival | Through completion of follow-up (estimated to be 10 years and 2 months)

CONTACTS AND LOCATIONS:
Overall Officials: Jiayi Huang, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu